CLINICAL TRIAL: NCT04020289
Title: A Randomized Controlled Trial of a Psychoeducational Program"BalancingMySwing" for Patients With Bipolar Disorder
Brief Title: A Psychoeducational Program "BalancingMySwing" for Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Esther Ching-Lan Lin, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU
Record Dates: First submitted 2019-07-08; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; depression; manic; illness perception
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania

STUDY DESIGN:
Intervention Model Description: Treatment as usual (TAU); and Psychoeducational Program "BalancingMySwing"
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "BalancingMySwing" (Experimental): Psychoeducational Program "BalancingMySwing" for bipolar disorder
  Interventions: Behavioral: Psychoeducational Program "BalancingMySwing"
- treatment as usual (TAU) (Other): Patients received treatment as usual
  Interventions: Behavioral: Psychoeducational Program "BalancingMySwing"

INTERVENTIONS:
Behavioral: Psychoeducational Program "BalancingMySwing" — Patients in the intervention arm will receive a nurse-lid 8-session psychoeducational 'BalancingMySwing" group psychotherapy

SUMMARY:
The psychoeducation BalancingMySwing (BMS) program has been developed manually and its feasibility has been tested in our previous study. This 3-year research project aimed to further examine the immediate and lasted effects of BMS program for BD, and to assess its knowledge dissemination and the transferability of its evidence-based practice across multiple sites.

DETAILED DESCRIPTION:
The psychoeducation BalancingMySwing (BMS) program has been developed manually and its feasibility has been tested in our previous study. This 3-year research project aimed to further examine the immediate and lasted effects of BMS program for bipolar disorders (BD), and to assess its knowledge dissemination and the transferability of its evidence-based practice across multiple sites.

During the first 2 years, a randomized controlled trial was conducted. Patients diagnosed with BD were recruited and 104 patients were randomly assigned to treatment as usual (TAU) or to 8 BMS sessions. A battery of three outcome indicators-social rhythm, illness perception, and symptom severity-were used to examine the effects of the two groups at baseline, after intervention, and every 3 months until half year. In addition, a pre- and post-test quasi-experimental study combined with qualitative design was used to assess the translational feasibility of BMS and to explore related barriers and facilitators of implementing BMS in clinical settings in the third year. Nurses from 4 Hospitals received the BMS training, and patients with BD received the BMS translated in practice were recruited.

ELIGIBILITY:
Inclusion Criteria:

* Had a DSM-IV(Diagnostic and Statistical Manual of Mental Disorders-IV) diagnosis of BP-I or II confirmed through the interviews using the Chinese version of the Modified Schedule of Affective Disorder and Schizophrenia-Lifetime.
* Able to speak and read Taiwanese or Taiwanese Mandarin Chinese
* Had signed a written consent form
* Agreed to accept the following medication therapy during the study: a mood stabilizer (valproic acid or lithium salts), an antidepressant, second generation antipsychotics, anxiolytics (lorazepam [< 8 mg/day]), and medicine to counteract side effects: extrapyramidal symptoms, tachycardia, and involuntary movement of smooth muscles in the gastrointestinal tract, urinary tract, lungs, etc.

Exclusion Criteria:

* Required immediate hospitalization
* Had any comorbidity with substance abuse or were current alcohol or drug abusers, or had been in the previous year
* Had been diagnosed with an organic psychosis, a neurodegenerative disease, a personality disorder, or impaired cognitive abilities

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Social Rhythm through Study Completion, at the 3rd and the 6th month after study completion | At baseline; through study completion, an average of 2 months; at the 3rd and the 6th month after study completion
  Social Rhythm Metric-5 items (SRM-5)-- The total scores range from 0 to 5; the higher the score the more regularly the activities occur.
Changes from Baseline Illness Perception through Study Completion, at the 3rd and the 6th month after study completion | At baseline; through study completion, an average of 2 months; at the 3rd and the 6th month after study completion
  Illness Perception Questionnaire-Revised (IPQ-R) has 3 subscales. The first subscale (identity) determines whether patients attribute specific symptoms to BD (total score: range = 0-10). The second subscale assesses 25 items of illness perceptions. The third subscale assessed the causes of BD. The second and third subscales are rated on a 5-point Likert scale (range: 1~5). A higher score on each item indicates a stronger belief in that illness perception.
Changes from Baseline Manic Symptom through Study Completion, at the 3rd and the 6th month after study completion | At baseline; through study completion, an average of 2 months; at the 3rd and the 6th month after study completion
  Young Mania Rating Scale (YMRS)--The total score of the 11-item YMRS is the summation of the 2 subscales (range: 0-60), and could be divided into four levels: 0 to 12 means remission, 13 to 19 means minimal severe, > 20 as diagnosed with mania based on DSM-IV(Diagnostic and Statistical Manual of Mental Disorders, IV) criteria, and over 25 showed obvious symptoms.
Changes from Baseline Depressive Symptom through Study Completion, at the 3rd and the 6th month after study completion | At baseline; through study completion, an average of 2 months; at the 3rd and the 6th month after study completion
  Hamilton Depression Rating Scale (HDRS)--The total score of the 17-item HDRS is the summation of the 2 subscales(ranged: 0- 52), and could be divided into four levels: 0-7 means remission, 8-13 means mild severe, 14-22 means moderate severe, and > 23 means very severe.

CONTACTS AND LOCATIONS:
Overall Officials: Esther C Lin, Principal Investigator — National Cheng Kung University

IPD SHARING:
Plan to Share IPD: Yes
We plan to use only for data analysis and publication without any recognized individual identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data analysis and publication will have occur at the end of the study, and continue after 7 months of the summary data are published.
Access Criteria: Only the research members in out research team can access individual participant data (IPD) and any additional supporting information and only for statistic data analysis and publication under the PI supervision. The PI will review all information shared to follow the research purpose.

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04020289/SAP_001.pdf